CLINICAL TRIAL: NCT05998681
Title: The Effects of Education on Breastfeeding and Basic Maternal-neonatal Care and Mobile Messaging on Breastfeeding and Motherhood Experience: A Randomized Controlled Trial
Brief Title: Effects of Education on Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra SABANCI BARANSEL, Assistant professor, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/3809
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Education; Mobile Messages; Breastfeeding Self-efficacy; Breastfeeding Attitude; Maternal Experience Satisfaction
Keywords: primipar; breastfeeding; education; self-efficacy; attitude; satisfaction
MeSH Terms: conditions — Breast Feeding; Behavior; Personal Satisfaction | interventions — Lactation

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial
Who Masked: Participant
Masking Description: This study was designed as a randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding and Basic Maternal-Neonatal Care and mobile messages group (Experimental): In the study, education on "Breastfeeding and Basic Maternal-Neonatal Care" was given to the women in the experimental group within the first 24 hours after the birth, and the training topics were sent as a mobile message for 6 weeks after the birth.
  Education on "Breastfeeding and Basic Maternal-Neonatal Care" was given in 2 postpartum sessions. In the first session, breastfeeding education was given to women in practice, together with the first postpartum breastfeeding. At the beginning of the second session, breastfeeding training was repeated and then Basic Maternal-Neonatal Care training was given. The first session was given at the first breastfeeding time, and the second session was given between 20-24 hours after birth. Each session lasted approximately 20-25 minutes. In order to solve the problems of the mothers, questions, and answers were made before discharge, and breastfeeding of the mothers was observed.
  Interventions: Other: Breastfeeding and Basic Maternal-Neonatal Care and mobile messages
- Routine checks (No Intervention): The researchers applied no initiative to the control group, and the women in the control group solely had the routine checks. The women in the control group filled out all pretest forms(A sociodemographic questionnaire including questions about age, educational level, employment, income level, whether the pregnancy was planned and the gender of the baby, as well as the personal phone numbers of the women, Breastfeeding Self-Efficacy Scale (BSES), IOWA-Infant Feeding Attitude Scale (IIFAS), and Being a Mother Scale (BaM-13) . The BSES, IIFAS, and BaM-13 were re-administered to all participants at postpartum 6 weeks as post-tests. In addition, the method by which the participants continued to feed their babies, their use of bottles or pacifiers, and their nipple problems were recorded in the form created by the researchers. Post-test data were collected by the researchers by contacting the participants by phone.

INTERVENTIONS:
Other: Breastfeeding and Basic Maternal-Neonatal Care and mobile messages — Participants in the experimental group were provided with education on "Breastfeeding and Basic Maternal-Neonatal Care" at the hospital and mobile messages were sent with the same content as education program for 6 weeks after discharge.
  Arms: Breastfeeding and Basic Maternal-Neonatal Care and mobile messages group

SUMMARY:
Objective: This study aims to investigate the effectiveness of education on breastfeeding and basic maternal-neonatal care and mobile message support given to primiparous women in the postpartum period on breastfeeding and motherhood experiences.

Methods: This prospective randomized controlled study was conducted in a hospital located in a city in Turkiye, with 130 primiparous patients in the postpartum period (65 individuals in the experimental group and 65 individuals in the control group). Participants in the experimental group were provided with education on "Breastfeeding and Basic Maternal-Neonatal Care" at the hospital and mobile messages were sent with the same content as education program for 6 weeks after discharge.

DETAILED DESCRIPTION:
Design This study was designed as a prospective randomized controlled study to determine the effectiveness of education on breastfeeding and basic maternal-neonatal care applied to primiparous women in the postpartum period and mobile messages on breastfeeding and motherhood experience.

Sample Inclusion criteria for this study were: (1) Primiparous; (2) aged ≥18 years; (3) having a healthy newborn; (4) participants who did not have an obstacle to postpartum breastfeeding and agreed to participate in the study were included in the study by simple random sampling method.

The study sample consisted of women hospitalized in the postpartum service of a hospital located in a province in eastern Turkey. In the postpartum service of the hospital, women who gave birth by vaginal or cesarean section are hospitalized. Early discharge procedures are performed after 24 hours for women who have had a vaginal delivery, and 48 hours for women who have had a cesarean delivery. Breastfeeding education is routinely provided in the hospital's postpartum service; however, the continuity and effectiveness of breastfeeding are not followed, and there is no information on neonatal care such as baby bathing, vaccination time, and training on emergencies that require a doctor's consultation.

Power analysis was performed using a web-based software to calculate the sample size for the research. The sample size was calculated as 65 for each group (65 participants in the experimental group and 65 participants in the control group) with a 5% error level, bidirectional significance level, 95% confidence interval, 80% ability to represent the population (power), and assuming that the Breastfeeding Self-Efficacy score which is 48.2 (standard deviation 7.7) will increase by 4 points.

Measures A questionnaire was created to determine the introductory characteristics of women and newborns and the breastfeeding process of women, and the Breastfeeding Self-Efficacy Scale (BSES), IOWA-Infant Feeding Attitude Scale (IIFAS), and Being a Mother Scale (BaM-13) were used to collect the data.

The BSES is a 33-item scale developed by Dennis and Faux in order to evaluate how competent mothers feel about breastfeeding. Later, in 2003, a 14-item short form of the scale was developed. The short form is easier to administer and accurately assesses breastfeeding self-efficacy. The BSES is a 5-point Likert-type scale, with each item rated from 1 (never sure) to 5 (always sure). The minimum score that can be obtained from the scale is 14, and the maximum score is 70. High scores indicate high breastfeeding self-efficacy. The Turkish adaptation of the scale was made by Tokat et al. and the Cronbach's alpha reliability coefficient was found to be 0.86.

The IIFAS aims to determine mothers' attitudes toward breastfeeding and to estimate the duration of breastfeeding. Cronbach's alpha reliability coefficient was determined as 0.71. The scale is a five-point Likert type and the number of items is 17. The total attitude score varies between 17 and 85, and a high score indicates a positive attitude toward breastfeeding.

The BaM-13 was developed by Matthey in 2011, and its Turkish validity and reliability study was conducted by Sevgi-Güler. The scale aims to determine mothers' experiences of motherhood. The scale, which consists of a total of 13 items, is a 4-point Likert-type scale and each item is scored between 0-3. The total score ranges from 0 to 39, and high scores on the scale indicate less satisfaction with the "motherhood" experience. The Cronbach's alpha reliability coefficient of the scale was determined as 0.76 .

Data Collection Data were collected between October 2022 and June 2023. The women assigned to the experimental and control groups were first informed about the study. Introductory characteristics such as age, educational level, employment, income level, whether the pregnancy was planned and the gender of the baby, as well as the personal phone numbers of the women, were recorded in the form created by the researchers. As pre-tests, the BSES, IIFAS, and BaM-13 were applied. The pre-test data were collected by the researchers using face-to-face interview method in the single rooms where the women stayed in the hospital.

The BSES, IIFAS, and BaM-13 were re-administered to all participants at postpartum 6 weeks as post-tests. In addition, the method by which the participants continued to feed their babies, their use of bottles or pacifiers, and their nipple problems were recorded in the form created by the researchers. Post-test data were collected by the researchers by contacting the participants by phone.

Intervention In the study, education on "Breastfeeding and Basic Maternal-Neonatal Care" was given to the women in the experimental group within the first 24 hours after the birth, and the training topics were sent as a mobile message for 6 weeks after the birth. Educational content and messages created by the researchers in line with the guidelines of ACOG and WHO, together with the literature review, were organized with the opinion of 5 experts who are experts in their field. The content of education and mobile messages were as follows: the importance of breastfeeding, breastfeeding techniques and things to be considered while breastfeeding, milking and storage conditions, nipple problems, postpartum mother-neonatal care, post-discharge emergencies.

Education on "Breastfeeding and Basic Maternal-Neonatal Care" was given to the participants individually by B.E., one of the expert researchers. In addition, mobile messages were also conveyed to the participants by B.E., one of the researchers. Education on "Breastfeeding and Basic Maternal-Neonatal Care" was given in 2 postpartum sessions. In the first session, breastfeeding education was given to women in practice, together with the first postpartum breastfeeding. At the beginning of the second session, breastfeeding training was repeated and then Basic Maternal-Neonatal Care training was given. The first session was given at the first breastfeeding time, and the second session was given between 20-24 hours after birth. Each session lasted approximately 20-25 minutes. In order to solve the problems of the mothers, questions, and answers were made before discharge, and breastfeeding of the mothers was observed. The trainings were given by the method of direct expression through brochures. Information messages were sent by the researcher via mobile message between 08:00 and 10:00 every day for 6 weeks following the 1st day after discharge. No intervention was applied to the women in the control group by the researcher. Breastfeeding training, which is included in the standard care of the hospital, was given to these women by the healthcare professionals in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Primiparous;
2. aged ≥18 years;
3. having a healthy newborn;
4. participants who did not have an obstacle to postpartum breastfeeding and agreed to participate in the study

Exclusion Criteria:

1. Unable to communicate in Turkish
2. Those with diagnosed psychological health problems will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women in the first 24 hours after the birth
Enrollment: 130 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale (BSES) | Change inbreastfeeding self-efficacy levels at 6 weeks
  The BSES is a 33-item scale developed by Dennis and Faux in order to evaluate how competent mothers feel about breastfeeding. Later, in 2003, a 14-item short form of the scale was developed. The short form is easier to administer and accurately assesses breastfeeding self-efficacy. The BSES is a 5-point Likert-type scale, with each item rated from 1 (never sure) to 5 (always sure). The minimum score that can be obtained from the scale is 14, and the maximum score is 70. High scores indicate high breastfeeding self-efficacy.

SECONDARY OUTCOMES:
IOWA-Infant Feeding Attitude Scale (IIFAS) | Change in attitudes towards breastfeeding at 6 weeks
  The IIFAS aims to determine mothers' attitudes toward breastfeeding and to estimate the duration of breastfeeding. Cronbach's alpha reliability coefficient was determined as 0.71. The scale is a five-point Likert type and the number of items is 17. The total attitude score varies between 17 and 85, and a high score indicates a positive attitude toward breastfeeding.
Being a Mother Scale (BaM-13) | Change in satisfaction with the "motherhood" experience levels at 6 weeks
  The BaM-13 was developed by Matthey in 2011, and its Turkish validity and reliability study was conducted by Sevgi-Güler. The scale aims to determine mothers' experiences of motherhood. The scale, which consists of a total of 13 items, is a 4-point Likert-type scale and each item is scored between 0-3. The total score ranges from 0 to 39, and high scores on the scale indicate less satisfaction with the "motherhood" experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Sabanci Baransel, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No